CLINICAL TRIAL: NCT00000510
Title: Platelet-Inhibitor Drug Trial in Coronary Angioplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 29; R01HL031025 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2005-03

CONDITIONS: Angina Pectoris; Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Angina Pectoris; Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Aspirin; Dipyridamole; Angioplasty, Balloon, Coronary

INTERVENTIONS:
Drug: aspirin
Drug: dipyridamole
Procedure: angioplasty, transluminal, percutaneous coronary

SUMMARY:
To determine the effectiveness of dipyridamole and aspirin in prevention of restenosis of the dilated lesion in patients who had undergone percutaneous transluminal coronary angioplasty (PTCA). Secondary aims were to determine the effectiveness of platelet inhibitor therapy in reducing the incidence of coronary events and the severity and incidence of angina.

DETAILED DESCRIPTION:
BACKGROUND:

By dilating coronary stenoses, PTCA can relieve angina pectoris and improve exercise tolerance and left ventricular function. However, restenosis occurs in 20-30 percent of dilated stenoses within three to six months following PTCA making it necessary to restrict patient activities, resume antianginal medications, repeat PTCA, or perform coronary artery bypass surgery.

Balloon dilatation of the atherosclerotic lesion damages the endothelium, intima, and media of the artery. This may lead to restenosis via platelet deposition, mural thrombus formation, and intimal proliferation by mechanisms that appear similar to those causing aortocoronary vein graft (ACVG) occlusions. It had been demonstrated that dipyridamole plus aspirin therapy suppressed these mechanisms of ACVG occlusion in the animal model, prolonged a shortened platelet survival in patients with coronary artery disease, and reduced ACVG occlusions in patients both early and late after the operation. Thus, a trial of these drugs in patients undergoing PTCA was a logical and necessary step to reduce the major shortcoming of the initially successful PTCA therapy, namely the high rate of restenosis.

DESIGN NARRATIVE:

Randomized, double-blind, fixed sample. Patients were randomized to treatment with dipyridamole plus aspirin or placebo.

The study completion date listed in this record was obtained from the Query/View/Report (QVR) System.

ELIGIBILITY:
Patients to age 80 with angina pectoris.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1983-09; Study Completion 1988-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Chesebro — Mayo Foundation